CLINICAL TRIAL: NCT07280832
Title: Open-Label, Multicenter Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of JMT108 Injection in Participants With Unresectable or Metastatic Melanoma
Brief Title: Phase I/II Clinical Study of JMT108 Injection for the Treatment of Advanced Malignant Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JMT108-003
Record Dates: First submitted 2025-11-28; First posted 2025-12-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Unresectable Locally Advanced or Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter Phase I/II clinical study
Masking Description: This is an open-label, multicenter Phase I/II clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase I: Dose Escalation Stage (Experimental): JMT108 intravenous (IV) administration, use as specified in the clinical study protocol.
  Interventions: Drug: JMT108
- Phase IIa: Dose Expansion Stage (Experimental): The administered dose of JMT108 selected by the SMC.
  Interventions: Drug: JMT108
- Phase IIb: Cohort 1 (Experimental): RP2D of JMT108 selected by the SMC.
  Interventions: Drug: JMT108
- Phase IIb: Cohort 2 (Experimental): RP2D of JMT108 selected by the SMC.
  Interventions: Drug: JMT108

INTERVENTIONS:
Drug: JMT108 — Intravenous (IV) administration

SUMMARY:
This is an open-label, multicenter Phase I/II clinical study conducted in participants with unresectable locally advanced or metastatic melanoma, aiming to evaluate the safety, tolerability, pharmacokinetic characteristics, and efficacy of JMT108 Injection in this population. The study consists of Phase I and Phase II (including Phase IIa and Phase IIb), where Phase I is the dose-escalation stage, Phase IIa is the dose-expansion stage, and Phase IIb is the cohort-expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old.
2. Histologically or cytologically confirmed unresectable locally advanced or metastatic melanoma.
3. Participants with unresectable locally advanced or metastatic melanoma who have failed prior standard treatment or have no available standard treatment will be enrolled in Phase I and Phase IIa; those who have received or not received prior standard treatment will be enrolled in Phase IIb.
4. According to the response evaluation criteria for solid tumors (RECIST 1.1), having at least one measurable lesion.
5. ECOG PS of 0-1.
6. Expected survival ≥ 3 months.
7. Participants with adequate organ functions.
8. Female and male patients of childbearing age agree to take adequate contraceptive measures during and upon completion of the study for 6 months after the last dose. Female participants of childbearing age must have a negative blood pregnancy test within 7 days before the first dose or randomization.
9. Voluntarily agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, or other unapproved clinical trial drugs or treatments within 4 weeks prior to the first administration of the study drug.
2. Prior use of IL-2/IL-15 cytokine therapy.
3. Received major organ surgery (excluding needle biopsy) or experienced severe trauma within 4 weeks prior to the first administration of the study drug, or requires elective surgery during the study period.
4. Received systemic glucocorticoids or other immunosuppressive therapy within 14 days prior to the first use of the study drug. Exceptions include the following situations: receiving physiological replacement doses of hydrocortisone or other equivalent doses of hormonal therapy (i.e., prednisone ≤ 10 mg/day or other equivalent doses of hormones); receiving topical, ophthalmic, intra-articular, intranasal, and inhaled glucocorticoid therapy; receiving short-course glucocorticoids for preventive treatment (e.g., prevention of contrast agent allergy).
5. Known active central nervous system (CNS) metastases and/or leptomeningeal metastases. Patients with stable brain metastases who do not require local treatment for brain metastases are eligible for inclusion.
6. Patients with active infections requiring intravenous anti-infective therapy within 14 days prior to the first administration.
7. Has a history of severe cardiovascular and cerebrovascular diseases.
8. Has active or recurrent autoimmune diseases.
9. Has a known history of receiving immunotherapy with the occurrence of grade ≥3 immune-related adverse events (irAEs) (excluding immune-related endocrine abnormalities that have been stabilized) or grade ≥2 immune-related myocarditis.
10. Has a history of arterial or venous thrombosis within 6 months prior to the first administration.
11. Has a history of serous effusions such as ascites or pleural effusion requiring drainage within 14 days prior to the first administration.
12. Has a history of other malignant tumors within 5 years prior to the first administration or concurrent other malignant tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) (Phase I) | Approximately 28 days.
  To evaluate the safery of JMT108 in subjects.
Adverse Events (AEs) (Phase I) | Through study completion, an average of 1 year
  To evaluate the safery of JMT108 in subjects.
Overall Response Rate (ORR) (Phase II) | To evaluate the efficacy of JMT108 in subjects.
  Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Through study completion, an average of 1 year.
  To evaluate the systemic pharmacokinetics of JMT108 in subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- BeiJing Cancer Hospital EC, Beijing, Beijing Municipality, China